CLINICAL TRIAL: NCT01809457
Title: Effectiveness of Educational Poster to Secondary Students Regarding Knowledge of Emergency Management of Dental Trauma - A Cluster Randomised Controlled Trial
Brief Title: Effectiveness of Dental Trauma Educational Poster to Secondary Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Cecilia Young, Principal investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: S01 / UW 11-177
Record Dates: First submitted 2013-03-10; First posted 2013-03-12 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Injuries
Keywords: educational poster, knowledge, dental trauma,
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- educational poster (Experimental): poster display for 2 weeks in classrooms,
  Interventions: Other: educational poster
- control (No Intervention): no intervention, waiting for two weeks

INTERVENTIONS:
Other: educational poster — educational poster for dental trauma
  Arms: educational poster

SUMMARY:
to investigate the effectiveness of the educational poster regarding knowledge of dental trauma for the secondary school students

DETAILED DESCRIPTION:
To investigate the effectiveness of the educational poster about dental trauma to increase the knowledge of secondary students.

Schools will be randomly divided into two groups, baseline score of knowledge in questionnaire will be collected for all subjects. Poster will be sent to intervention group, the school will place it at the notice broad or area of similar function in the classroom. For the control group, nothing will be given, then after 2 weeks, the score of knowledge by the second questionnaire of both groups will be collected again.

To compare the difference in knowledge before and after in both groups, statistical test will be performed.

Investigators conduct a cluster randomized controlled trial. A list of secondary schools was requested from the Education Bureau. Secondary schools will be invited to join the study and then randomized to the intervention group and the control group in the unit of school using computer generated numbers. All students will fill in the first questionnaire and send it back to the investigator in 1 week. Then copies of the same poster will be given to the intervention schools, these schools will be requested to place them in the classrooms of the participating students. No poster will be given to the control group. After 2 weeks, the poster will be removed. The same questionnaire will be filled out by all the students in both groups and sent back in 1 week. Then the data will be processed to show whether the poster is effective to improve the knowledge of the students.

ELIGIBILITY:
Inclusion Criteria

- All secondary schools in Hong Kong that the students can read Chinese or English

Exclusion Criteria

- no school consent or individual guardian consent

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 671 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
knowledge score | 2 weeks
  a questionnaire to test the knowledge score

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Young, BDS, MPH, Principal Investigator — Independent
Locations (1):
- secondary schools in Hong Kong, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Young C, Wong KY, Cheung LK. Effectiveness of educational poster on knowledge of emergency management of dental trauma--part 2: cluster randomised controlled trial for secondary school students. PLoS One. 2014 Aug 5;9(8):e101972. doi: 10.1371/journal.pone.0101972. eCollection 2014. PMID 25093728